CLINICAL TRIAL: NCT02055573
Title: Can we Promote Early Literacy and Prevent Shaken Baby Syndrome in the Well Child Nursery?.A Randomized Controlled Study, The Early ABC Study.
Brief Title: The Early ABCs Study
Acronym: EarlyABCs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: Lifespan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: WIH 13-0080
Record Dates: First submitted 2014-01-10; First posted 2014-02-05 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Abusive Head Trauma; Early Literacy
Keywords: Abusive Head Trauma; Early Literacy; Parental Education; Low Income
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ready To Learn (Experimental): 1) The Ready to Learn (RTL) arm will receive a DVD in both Spanish and English and a bilingual booklet (both produced by Parents' action for Children) addressing the benefits of reading, talking and playing with young children, as well as a new children's board book.
  Interventions: Other: Ready To Learn (RTL)
- All Babies Cry (Experimental): 2) The All Babies Cry (ABC) arm will receive a DVD in both, Spanish and English and a bilingual booklet (both produced by VIDA Health Communications, INC) explaining crying as part of normal infant behavior, highlighting signs of parental distress and providing strategies to sooth parents and their children
  Interventions: Other: All Babies Cry (ABC)

INTERVENTIONS:
Other: Ready To Learn (RTL) — See arm description
  Arms: Ready To Learn
Other: All Babies Cry (ABC) — See arm description
  Arms: All Babies Cry

SUMMARY:
Regular reading with young children strengthens the parent-child relationship and builds their language, literacy and social emotional skills. Parent knowledge of normal variation of infant crying and of the dangers of shaking a baby as well as their ability to cope with infant irritability are likely factors in their successful adjustment to parenthood and the prevention of this tragic act.

Purpose: Identify easily implementable interventions for economically disadvantaged mothers in the newborn period which 1) Promote early literacy behaviors and early nurturing parent-child relationships and 2) Increase mother's knowledge of normal crying patterns, the dangers of shaking a baby and her ability to cope with parenting stresses.

Design/Methods: A convenience sample of 300 low income (insured by Medicaid) new mothers of healthy singleton, full term infants in the level 1 mother/baby unit at Women & Infants Hospital will be invited to participate in a Randomized Controlled Trial study of educational videos and materials for parents. They will be randomized into one of two intervention groups. 1) The Ready to Learn (RTL) arm will receive a DVD in both Spanish and English and a bilingual booklet (both produced by Parents' action for Children) addressing the benefits of reading, talking and playing with young children, as well as a new children's board book. 2) The All Babies Cry (ABC) arm will receive a DVD in both, Spanish and English and a bilingual booklet (both produced by VIDA) explaining crying as part of normal infant behavior, highlighting signs of parental distress and providing strategies to sooth parents and their children. We will enroll 75 mothers who speak Spanish primarily at home in each intervention group, as well as 75 mothers who speak primarily English. The RTL mothers will serve as controls for the ABC mothers and vice versa. Before reviewing the materials, mothers will be asked to respond to a baseline interview with socio-demographic information, questions regarding Early Literacy promotion, reading with children and their own reading habits as well as general knowledge on the prevention of shaking a baby and handling their own stress. Follow up phone interviews will be conducted by a bilingual research assistant blind to the intervention status at 2-5 months post-partum containing similar questions. Consenting mothers will receive a bag of diapers at the completion of enrollment interview as an incentive for participating in the study. Data will be entered into Excel and transferred into STATA for analysis. Frequency counts will be generated for demographic, literacy related and parental knowledge and stress variables in the two intervention arms. Chi-Square and T-tests will be used to compare literacy and parental knowledge outcomes for each intervention group at both follow up interviews.

Hypotheses: 1) Mothers in the RTL branch will recognize the importance of reading to their babies, initiating this activity at earlier ages and reading more often with them. 2) Mothers in the ABC branch will gain an understanding of crying as part of normal infant behavior and build strategies to sooth themselves and their newborns.

DETAILED DESCRIPTION:
Quality assurance Plan: The PI and collaborators will be overseen collection and processing of data.

Standard Operating Procedures:

Recruitment: A bilingual Research Assistant will review mother's records at Women & Infants' Hospital mother-baby unit to identify eligible mothers.

Dyads will be excluded if the mother:

* Is not insured by Medicaid, Ritecare, or Neighborhood Health Plan.
* Is not fluent in either English or Spanish.
* Is younger than 18 years of age.
* Will not be taking the baby home at hospital discharge.
* Will be leaving USA within the following 6 months for longer than two weeks.
* Is discharged from the hospital prior to being approached or scheduling interview.
* Does not have access to DVD player
* Refuses to participate in the study.

Dyads will be excluded if the infant:

* Is born premature (<37 wks G.A)
* Is born at low birth weight (<5 pounds or 2500 grams at birth)
* Spent >24 hours in the Neonatal Intensive Care Unit
* Was born with a significant anomaly or genetic syndrome associated with delay
* Has a P.R.E with a hold with DCYF

Data Collection/Management and Analysis:

A convenience sample of 300 low income (insured by Medicaid) new mothers of healthy singleton, full term infants in the level 1 mother/baby unit at Women & Infants Hospital will be invited to participate in a Randomized Controlled Trial of educational videos and materials for parents. They will be randomized into one of two intervention groups. 1) The Ready to Learn (RTL) arm will receive a DVD in both Spanish and English and a bilingual booklet (both produced by Parents' action for Children) addressing the benefits of reading, talking and playing with young children, as well as a new children's board book. 2) The All Babies Cry (ABC) arm will receive a DVD in both, Spanish and English and a bilingual booklet (both produced by VIDA Health Communications, INC) explaining crying as part of normal infant behavior, highlighting signs of parental distress and providing strategies to sooth parents and their children. We will enroll 75 mothers who speak Spanish primarily at home in each intervention group, as well as 75 mothers who speak primarily English in each arm. The RTL mothers will serve as controls for the ABC mothers and vice versa. Before reviewing the materials, mothers will be asked to respond to a baseline interview with socio-demographic information, questions regarding Early Literacy promotion, reading with children and their own reading habits as well as general knowledge on the prevention of shaking a baby and handling their own stress. Follow up phone interviews will be conducted by a bilingual research assistant blinded to the intervention status at 2-5 months post-partum containing similar questions. Data will be entered into Excel and transferred into STATA for analysis.

Sample Size calculation:

For power analysis, we used categorical (behavioral) outcomes to arrive at conservative estimates of sample sizes with a 0.05 significance level. Effect sizes for differences in proportions are based on Cohen's h statistic (Cohen, 1988), computed for 80% power and Two-tailed significance test at alpha = 0.05 with equal numbers of participants in the intervention and control groups and a Confidence Interval of 95%.

From a previous study of the All Babies Cry intervention at 5 weeks postpartum 36% of control group answered similar knowledge questions correctly, compared to 47% of those receiving the All Babies Cry Intervention. This resulted in a difference of 11% and SD of 18 in the control group and 19 in the intervention group.

Based on this using Open Epi for sample size calculation we arrived at a group size of 45 subjects in each branch of the study. Althouhg in the original All Babies Cry Intervention we had a follow up rate of 77% at 17 weeks, our current estimates are closer to 40-45%. To account for a possible loss to follow up of 60% of subjects we will increase the sample size from 45 to 75 individuals in each group for a total of 150 subjects in each branch of the study.

Previous studies of Early Literacy interventions in low income families have shown larger differences in similar literacy outcomes to ours. We are therefore basing our calculations on a more conservative data assumption.

Statistical Analysis:

Frequency counts will be generated for demographic, literacy related and parental knowledge and stress variables in the two intervention arms. Chi-Square and T-tests will be used to compare literacy and parental knowledge outcomes for each intervention group at baseline and at both follow up interviews.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of healthy Singleton, full term infants
* Born at Women & Infants Hospital

Exclusion Criteria:

Mothers will be excluded if they:

* Are not insured by Medicaid, Ritecare, or Neighborhood Health Plan.
* Are not fluent in either English or Spanish.
* Are younger than 18 years of age.
* Will not be taking the baby home at hospital discharge.
* Will be leaving USA within the following 6 months for longer than two weeks.
* Is discharged from the hospital prior to being approached or scheduling interview.
* Do not have access to DVD player
* Refuse to participate in the study.

Mothers will be excluded if the infant:

* Is born premature (<37 wks G.A)
* Is born at low birth weight (<5 pounds at birth or 2500 grams)
* Spent >24 hours in the Neonatal Intensive Care Unit
* Was born with a significant anomaly or genetic syndrome associated with delay
* Has a P.R.E with a hold with DCYF

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Days/week mothers report reading with their infants | 2-5 months
  Mothers are asked how many days/week they read with their babies at 2-5 months. We hypothesize that mothers in the RTL Arm will report that they read with their babies more days/week compared to ABC Arm mothers.
Reading with their baby is one of mother's favorite shared activities | 2-5 months
  Mothers are asked what their 3 favorite things to do with their babies are. We hypothesize that more mothers in the RTL Arm will spontaneously mention reading books together.
Knowledge of the typical peak of infant crying | 2-5 months
  At follow-up interview mothers are asked if they know at what age infants tend to cry the most and they are given 7 options. We hypothesize that more mothers in the ABC Arm of the study will correctly identify 6-8 weeks as the peak of infant crying compared to RTL Arm mothers.
Having heard what can happen if a baby is shaken | 2-5 months
  At follow-up mothers are asked if they have heard or read what could happen if a baby is shaken. We hypothesize that more mothers in the ABC arm of the study will report having heard of what could happen if a baby is shaken.

SECONDARY OUTCOMES:
Reading together is one of the baby's 3 favorite activities. | 2-5 months
  At follow-up, mothers are asked what their baby's 3 favorite things to do are. We hypothesize that more mothers in the RTL Arm will spontaneously mention reading books with their parents as one of the baby's 3 favorite activities, compared to ABC arm mothers.
Number of children's books in the home | 2-5 months
  At follow-up mothers are asked how many children's books are in their home. We hypothesize that mothers in the RTL arm will report having more children's books in their homes compared to the numbers of children's books in the homes of ABC arm mothers.
Reading with their baby is identified as a way of preparing him/her for school | 2-5 months
  Mothers are asked if there is anything they plan to do with their child to help the child do well when he/she goes to school. We hypothesize that more RTL mothers compared to ABC mothers will spontaneously mention reading together or books as a way of promoting their child's readiness for school.
Talking, singing and/or playing with their babies is identified as a favorite shared activity | 2-5 months
  Mothers are asked what their 3 favorite things to do with their babies are. We hypothesize that more mothers in the RTL Arm will spontaneously mention talking, singing and/or playing together as a favorite shared activity compared to ABC Arm mothers.
Number of calming strategies for parenting stress identified | 2-5 months
  At follow-up mothers are asked to identify ways of calming themselves if their baby is crying inconsolably. We hypothesize that mothers in the ABC arm will identify more strategies for calming themselves if their baby is crying, compared to RTL arm mothers.
Number of soothing strategies to calm fussy babies identified | 2-5 months
  At follow-up mothers are asked to identify ways of soothing their babies if they are crying inconsolably. We hypothesize that mothers in the ABC arm will identify more strategies for soothing their babies if they are crying inconsolably, compared to RTL arm mothers.
Knowledge that responding to babies younger than 6 months of age whenever they cry won't spoil them | 2-5 months
  At follow-up interview mothers are asked if they believe that by responding to a baby in the first 6 months of life every time he/she starts to cry he/she can get spoiled. We hypothesize that more mothers in the ABC Arm of the study will know that they can't spoil a baby less than 6 months old by responding to all their cries, as compared to RTL arm mothers.
Knowledge that shaking a baby can cause brain damage or death | 2-5 months
  At follow-up interview mothers are asked if they have heard what could happen if a baby is shaken. We hypothesize that more mothers in the ABC Arm of the study will correctly identify that babies can sustain brain damage or die if they are shaken compared to RTL Arm mothers

OTHER OUTCOMES:
Other caregivers are reading with baby | 2-5 months
  Mothers will be asked who if anyone else reads with their baby?. We hypothesize that mothers in the RTL arm will be more likely to report that someone else reads with their baby as compared to mothers in the ABC arm
DVD/Booklet promotes reading, playing or talking with baby | 2-5 months
  At follow up interview mothers will be asked which parts of the DVD/Booklet they found helpful?. We hypothesize that RTL arm mothers will be more likely to report guidance around reading, playing or talking with baby was helpful compared to ABC arm mothers
DVD/Booklet teaches how to calm baby or self | 2-5 months
  At follow up interview mothers will be asked which parts of the DVD/Booklet they found helpful?. We hypothesize that ABC arm mothers will be more likely to report guidance around how to sooth a baby and/or handle parenting stress was helpful compared to RTL arm mothers

CONTACTS AND LOCATIONS:
Overall Officials: Marcia W VanVleet, MD, MPH, Principal Investigator — Women & Infants' Hospital
Locations (1):
- Women & Infants' Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Background] Garner AS, Shonkoff JP; Committee on Psychosocial Aspects of Child and Family Health; Committee on Early Childhood, Adoption, and Dependent Care; Section on Developmental and Behavioral Pediatrics. Early childhood adversity, toxic stress, and the role of the pediatrician: translating developmental science into lifelong health. Pediatrics. 2012 Jan;129(1):e224-31. doi: 10.1542/peds.2011-2662. Epub 2011 Dec 26. PMID 22201148
- [Background] Barr RG, Barr M, Fujiwara T, Conway J, Catherine N, Brant R. Do educational materials change knowledge and behaviour about crying and shaken baby syndrome? A randomized controlled trial. CMAJ. 2009 Mar 31;180(7):727-33. doi: 10.1503/cmaj.081419. Epub 2009 Mar 2. PMID 19255065
- [Background] Duursma E, Augustyn M, Zuckerman B. Reading aloud to children: the evidence. Arch Dis Child. 2008 Jul;93(7):554-7. doi: 10.1136/adc.2006.106336. Epub 2008 May 13. No abstract available. PMID 18477693
- [Background] Keeton CP, Perry-Jenkins M, Sayer AG. Sense of control predicts depressive and anxious symptoms across the transition to parenthood. J Fam Psychol. 2008 Apr;22(2):212-21. doi: 10.1037/0893-3200.22.2.212. PMID 18410208
- [Background] Lewin L. Shaken baby syndrome: facts, education, and advocacy. Nurs Womens Health. 2008 Jun;12(3):235-9. doi: 10.1111/j.1751-486X.2008.00328.x. No abstract available. PMID 18557853
- [Background] Lee C, Barr RG, Catherine N, Wicks A. Age-related incidence of publicly reported shaken baby syndrome cases: is crying a trigger for shaking? J Dev Behav Pediatr. 2007 Aug;28(4):288-93. doi: 10.1097/DBP.0b013e3180327b55. PMID 17700080
- [Background] Berkule SB, Dreyer BP, Huberman HS, Fierman AH, Mendelsohn AL. Attitudes about shared reading among at-risk mothers of newborn babies. Ambul Pediatr. 2007 Jan-Feb;7(1):45-50. doi: 10.1016/j.ambp.2006.10.004. PMID 17261482
- [Background] Evanoo G. Infant crying: a clinical conundrum. J Pediatr Health Care. 2007 Sep-Oct;21(5):333-8. doi: 10.1016/j.pedhc.2007.06.014. No abstract available. PMID 17825733
- [Background] Tomopoulos S, Dreyer BP, Tamis-LeMonda C, Flynn V, Rovira I, Tineo W, Mendelsohn AL. Books, toys, parent-child interaction, and development in young Latino children. Ambul Pediatr. 2006 Mar-Apr;6(2):72-8. doi: 10.1016/j.ambp.2005.10.001. PMID 16530142
- [Background] High PC, LaGasse L, Becker S, Ahlgren I, Gardner A. Literacy promotion in primary care pediatrics: can we make a difference? Pediatrics. 2000 Apr;105(4 Pt 2):927-34. PMID 10742349
- [Background] Golova N, Alario AJ, Vivier PM, Rodriguez M, High PC. Literacy promotion for Hispanic families in a primary care setting: a randomized, controlled trial. Pediatrics. 1999 May;103(5 Pt 1):993-7. doi: 10.1542/peds.103.5.993. PMID 10224178
- [Background] Barr RG. The normal crying curve: what do we really know? Dev Med Child Neurol. 1990 Apr;32(4):356-62. doi: 10.1111/j.1469-8749.1990.tb16949.x. No abstract available. PMID 2332126
- [Background] Mendelsohn AL, Mogilner LN, Dreyer BP, Forman JA, Weinstein SC, Broderick M, Cheng KJ, Magloire T, Moore T, Napier C. The impact of a clinic-based literacy intervention on language development in inner-city preschool children. Pediatrics. 2001 Jan;107(1):130-4. doi: 10.1542/peds.107.1.130. PMID 11134446
- [Background] Needlman R, Toker KH, Dreyer BP, Klass P, Mendelsohn AL. Effectiveness of a primary care intervention to support reading aloud: a multicenter evaluation. Ambul Pediatr. 2005 Jul-Aug;5(4):209-15. doi: 10.1367/A04-110R.1. PMID 16026185
- See also: 4. National Institute for Literacy. 2008. Developing early literacy: Report of the National Early Literacy Panel. — http://lincs.ed.gov/publications/pdf/NELPReport09.pdf